CLINICAL TRIAL: NCT02605850
Title: Effects of Phytonutrients on Vascular Health
Acronym: PomPAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB#15-001605
Record Dates: First submitted 2015-10-12; First posted 2015-11-16 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Cardiovascular Diseases
Keywords: heart health
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Water; pomegranate fruit rind

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ground beef patty + Water (Placebo Comparator): 32 healthy subjects, ages 18-35 years who meet all the eligibility criteria in the screening phase of the study will receive the ground beef patty + water to evaluate the clinical efficacy of pomegranate on vascular health.Then subjects will be randomized to consume pomegranate juice or extract. At visit 2, subjects will be tested before and after meal with pomegranate juice or extract, then take pomegranate product daily for 4 weeks. At visit 3, subjects will tested before and after test meal with pomegranate products.
  Interventions: Other: Water
- Ground beef patty + Pomegranate Extract (Active Comparator): 32 healthy subjects, ages 18-35 years who meet all the eligibility criteria in the screening phase of the study will receive the ground beef patty + water to evaluate the clinical efficacy of pomegranate on vascular health.Then subjects will be randomized to consume pomegranate juice or extract. At visit 2, subjects will be tested before and after meal with pomegranate juice or extract, then take pomegranate product daily for 4 weeks. At visit 3, subjects will tested before and after test meal with pomegranate products.
  Interventions: Dietary Supplement: Pomegranate extract
- Ground beef patty + Pomegranate Juice (Active Comparator): 32 healthy subjects, ages 18-35 years who meet all the eligibility criteria in the screening phase of the study will receive the ground beef patty + water to evaluate the clinical efficacy of pomegranate on vascular health.Then subjects will be randomized to consume pomegranate juice or extract. At visit 2, subjects will be tested before and after meal with pomegranate juice or extract, then take pomegranate product daily for 4 weeks. At visit 3, subjects will tested before and after test meal with pomegranate products.
  Interventions: Dietary Supplement: Pomegranate Juice

INTERVENTIONS:
Other: Water — All subjects will consume ground beef patty meal with water at the baseline visit.
  Arms: Ground beef patty + Water
Dietary Supplement: Pomegranate Juice — Pomegranate Juice will be taken 1/day for 4 weeks.
  Other Names: PJ
  Arms: Ground beef patty + Pomegranate Juice
Dietary Supplement: Pomegranate extract — Pomegranate extract will be taken 1/day for 4 weeks.
  Other Names: PomX
  Arms: Ground beef patty + Pomegranate Extract

SUMMARY:
This study will determine the effects of beneficial compounds of plant foods, such as pomegranate on cardiovascular health. This will be tested by asking healthy males to eat a high fat ground beef patty with pomegranate juice (PJ), pomegranate extract (PomX) or water and then measuring blood vessel dilation (endothelial function) by blood flow We also will measure the amount of Nitric Oxide (NO) in your blood and urine samples and sugar and insulin in blood. Healthy men have been chosen for this study because eating high fat hamburger patties can easily mimic in them the condition that causes atherosclerosis. The results from this study may help to explain how high fat foods can be harmful to the body and how beneficial plant foods can have on cardiovascular function

DETAILED DESCRIPTION:
A. Specific Aims and Objectives

1. Peripheral arterial reactivity by tonometry after a high fat meal with pomegranate consumption
2. To measure nitric oxide and insulin response after a high fat meal and pomegranate consumption These studies will lead to a better understanding of the role of bioactive substances from plant foods such as the pomegranate may demonstrate the importance of plant-based nutrients on cardiovascular health.

B. Background Polyphenols belong to the largest group of secondary metabolites produced by plants, mainly, in response to biotic or abiotic stresses such as infections, wounding, UV irradiation, exposure to ozone, pollutants, and other hostile environmental conditions. It is thought that the molecular basis for the protective action of polyphenols in plants is their antioxidant and free radical scavenging properties.

Pomegranate (Punica granatum L.) is grown commercially in the Near East, India, Spain, Israel and the United States (California) where it is of significant economic importance. Pomegranate fruits and products, including juice, tea, wine and extracts are widely consumed and recognized for their health benefits. Pomegranate (Punica granatum L.) fruit possesses strong antioxidant, anti-inflammatory and antiproliferative properties.

High-calorie meals rich in saturated fat can lead to transient exaggerated elevations in blood glucose, free fatty acids, and triglycerides. This condition, termed postprandial dysmetabolism, generates excess free radicals (or reactive oxygen species). The ensuing oxidative stress triggers a biochemical cascade throughout the circulation, inducing inflammation, and endothelial dysfunction. These postprandial changes, when repeated multiple times each day, can create a milieu conducive for the development of atherosclerotic risk factors and coronary heart disease (CHD).

In order to investigate the impact of pomegranate polyphenols on postprandial flow-mediated dilation, nitric oxide, glucose, insulin, triglycerides levels in men, we propose to achieve the following specific aims using a randomized study design:

1. Peripheral arterial reactivity by tonometry after a high fat meal with pomegranate consumption
2. To measure nitric oxide and insulin response after a high fat meal and pomegranate consumption

ELIGIBILITY:
Inclusion Criteria:

* 18 - 35 years old males (inclusive)
* Non-smokers
* Must weigh a minimum of 110 pounds
* Willing to maintain normal activity and eating patterns for the duration of the study
* Willing to maintain their normal diet for the duration of the study but avoid pomegranate products and ellagitannin rich foods.

Exclusion Criteria:

* Any chronic medical conditions
* Abnormal liver function (AST and ALT > 2 x upper limit)
* Currently taking steroidal drugs
* Cancer treated within the past two years
* Participation in a therapeutic research study within 30 days of baseline
* Use of antibiotics within one month
* Regular use of probiotics
* Allergy or sensitivity to pomegranate products
* Follow a vegetarian diet
* Known HIV positive

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Abnormal PAT Values That Are Related to Treatment | Change from Baseline vascular function at 6 weeks
  The major outcomes are PAT changes after a test meal with and without pomegranate.

SECONDARY OUTCOMES:
Number of Participants With Abnormal Laboratory Values That Are Related to Treatment | Change from Baseline laboratory values at 6 weeks
  Correlation between outcomes measures (e.g. between nitric oxide and insulin response) with mixed effects models.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.

REFERENCES:
- [Background] Ross R. The pathogenesis of atherosclerosis: a perspective for the 1990s. Nature. 1993 Apr 29;362(6423):801-9. doi: 10.1038/362801a0. PMID 8479518
- [Background] Bonetti PO, Lerman LO, Lerman A. Endothelial dysfunction: a marker of atherosclerotic risk. Arterioscler Thromb Vasc Biol. 2003 Feb 1;23(2):168-75. doi: 10.1161/01.atv.0000051384.43104.fc. PMID 12588755
- [Background] Kasprzak JD, Klosinska M, Drozdz J. Clinical aspects of assessment of endothelial function. Pharmacol Rep. 2006;58 Suppl:33-40. PMID 17332669
- [Background] Anderson TJ, Gerhard MD, Meredith IT, Charbonneau F, Delagrange D, Creager MA, Selwyn AP, Ganz P. Systemic nature of endothelial dysfunction in atherosclerosis. Am J Cardiol. 1995 Feb 23;75(6):71B-74B. doi: 10.1016/0002-9149(95)80017-m. PMID 7863979
- [Background] Nohria A, Gerhard-Herman M, Creager MA, Hurley S, Mitra D, Ganz P. Role of nitric oxide in the regulation of digital pulse volume amplitude in humans. J Appl Physiol (1985). 2006 Aug;101(2):545-8. doi: 10.1152/japplphysiol.01285.2005. Epub 2006 Apr 13. PMID 16614356
- [Background] Bonetti PO, Barsness GW, Keelan PC, Schnell TI, Pumper GM, Kuvin JT, Schnall RP, Holmes DR, Higano ST, Lerman A. Enhanced external counterpulsation improves endothelial function in patients with symptomatic coronary artery disease. J Am Coll Cardiol. 2003 May 21;41(10):1761-8. doi: 10.1016/s0735-1097(03)00329-2. PMID 12767662